CLINICAL TRIAL: NCT03443895
Title: A Phase 1, Single Center, Double-blind, Placebo-Controlled, Dose Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Effects of Multiple Oral Doses of AEF0117 in Healthy Male and Female Subjects
Brief Title: Multiple Ascending Dose to Study the Safety, Tolerability, PK and PD Effects of AEF0117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AEF0117-102; R01DA038875 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2018-02-23 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. Subjects and investigator will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: AEF0117 (Active Comparator): Subjects in cohorts 1 through 3 receive active treatments. Subjects in Cohorts 1 through 3 will receive a single dose of 0.6, 2 and 6mg respectively of AEF0117 on Day 1 to Day 7.
  Interventions: Drug: AEF0117 oral capsule
- Placebo (Placebo Comparator): Subjects in Cohorts1 through 3 will be randomly assigned in an 6:2 allocation to receive active or placebo treatments.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: AEF0117 oral capsule — 0.6, 2 and 6mg of AEF0117
  Arms: Experimental: AEF0117
Drug: Placebo oral capsule — Matching placebo capsule
  Arms: Placebo

SUMMARY:
The study is designated to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of escalating multiple oral doses of AEF0117 in healthy adult male and female subjects.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of escalating multiple oral doses of AEF0117. This will be a single center study in healthy male and female subjects. The study design will be a double-blind, randomized, placebo-controlled, single period, parallel group, multiple dose escalation with AEF0117.

Three dose levels are planned for the study with 8 subjects (6 active and 2 placebo) per dose level:

Dose Level I - 0.6 mg multiple oral dose of AEF0117 given on the morning of Day 1 to Day 7 Dose Level II - 2 mg multiple oral dose of AEF0117 given on the morning of Day 1 to Day 7 Dose Level III - 6 mg multiple oral dose of AEF0117 given on the morning of Day 1 to Day 7

The planned dose escalation schema may be amended based on the emerging PK and safety data, and an additional cohort may be added. Smaller dose escalation increments can also be implemented based on safety and PK results of previous dose levels. Each subject will participate in only one dose group.

Administration of AEF0117 to each dose cohort should not occur before participants in the previous dose cohort have been treated and data i.e. safety results and PK from those participants are reviewed in accordance with the protocol. Eligible subjects will be admitted to the research clinic at midday prior to dosing (Day -1) and remain in house until Day 14. Subsequently subjects will return to the research facility on an outpatient basis to have PK and safety assessments at 216 and 264 hours (Day 16 and Day 18) after the last dose (Day 7). PK samples and safety assessments will be done pre-dose and at different times post-dose.

Randomized subjects will receive a single oral dose per day on Days 1 through 7. Serial PK and PD blood samples and urine PK collections will be performed for 24 hours after the first dose administration (Day 1). Pre-dose PK and PD blood samples will then be obtained on Days 3, 4, 5 and 6 prior to the daily dose administration. Serial PK and PD blood samples and urine collections will be also performed for 48 hours after the last dose (Day 7), and blood samples will be obtained at 72, 96, 120, 144, 168, 216 and 264 hours after the last dose (Day 7).

Safety monitoring (physical examinations, vital sign measurement, 12 lead ECGs, clinical safety laboratory tests, and adverse event monitoring) will be performed throughout the study. Psychometrics tests (Bond & Lader VAS, ARCI, POMS) will be performed on D1 and D7 at pre-dose, tmax and 24 hours post-dose. CSSRS test will be performed at pre-dose of D1 and at D8. tmax will be determine according to PK results obtained in the AEF0117-101 clinical study. Subjects will have a final follow up/Study termination safety evaluation on Day 18.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy, non-smoking or smoking (<10 cigarettes per day) male of any race, at least 18 years old and no more than 55 years old, inclusive. As the effect of the study drug on sperm is still unknown, male subjects should refrain from donating sperm or plan a pregnancy with their partner throughout the study and after 90 days, and must report immediately to the study doctor if its partner becomes pregnant during the study and after 90 days. The male subject will have to use double-barrier contraceptive methods: male condoms and spermicide.
2. Be a healthy, non-smoking or smoking (<10 cigarettes per day) female of non-child-bearing potential between 18 years of age and 55 years of age, inclusive. Females may be accepted if they are documented to be surgically sterile (e.g., hysterectomy, tubal ligation) or post-menopausal [amenorrhea >1 year and FSH >25.8mlU/mL, cut off from Labcorp] with a negative pregnancy test. At least 30% of female.
3. Have a body weight ≥50 kg, with a body mass index (BMI) calculated as weight in kg/(height in m)2 from 18 to 30 kg/m2 (inclusive) at screening.
4. Have no significant diseases in the medical history and no clinically significant findings on physical examination including ECG, BP, HR, RR, temperature, C-SSRS test. Routine laboratory values should be within normal ranges or considered as NCS by the investigator. The Non Clinical Significant nature of the deviation will result from the integration of a full clinical examination with physical examination and lab tests in that contest by a certified physician.
5. Be informed of the nature of the study and provide written informed consent.
6. Be legally competent and able to communicate effectively with study personnel.

Exclusion Criteria:

1. Allergies to the Investigational Medicinal Product (IMP) or placebo and its excipients and known allergies to pregnenolone or its matching placebo or its ingredient
2. Acute signs of intoxication at screening or baseline assessment due to opiates or any type of stimulants, causing cognitive impairments
3. Severe learning disability, brain damage or pervasive developmental disorder ( as this may affect one of the end point that is being targeted)
4. Any disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems.
5. Have abnormal baseline values for the steroid hormones: cortisol, testosterone, estradiol and progesterone in accordance to their reproductive status (for example but not limited to surgical sterile or post-menopausal).
6. A history of alcoholism or drug addiction within the past 2 years, recent use (in the last month) of any recreational drugs, or positive results from a urine screen for substances of abuse or positive alcohol test.
7. A history of or current serious mental illness including active or recent suicidal ideation, severe psychological distress (e.g., active suicidal plans, psychosis, debilitating panic disorder) or/and an abnormal C-SSRS result.
8. A history of difficulty donating blood or inadequate venous access.
9. The donation of blood or plasma within 30 days prior to receiving study medication or received any blood and plasma for medical/surgical reasons or intention to donate blood or plasma within one month after receiving the study drug.
10. A positive hepatitis screen that tests for both hepatitis B surface antigen (HBsAg) and antibody to hepatitis C (HCV).
11. A positive test result for HIV antibody by enzyme immunoassay which is confirmed by Western immunoblot.
12. Ingestion of an investigational drug or product, or participation in a drug study within a period of 30 days prior to receiving study medication (for investigational drugs with an elimination half-life greater than 10 days, this will be extended to 60 days).
13. Use of any prescription or over-the-counter (OTC) drug therapy, including herbal, homeopathic, vitamins, minerals and nutritional supplements, bodybuilding supplements unapproved by the sponsor, within 2 weeks prior to receiving the study medication (for drugs with an elimination half-life greater than 10 days, this will be extended to 60 days). The use of any food supplement or body cream containing pregnenolone or any other steroid including phytosteroids.
14. Use of a drug therapy known to induce or inhibit hepatic drug metabolism within 30 days prior to receiving study medication or during the study.
15. Use of psychoactive and/or psychotropic medication (including sedative, antidepressant and antipsychotics), or medication that alters the hypothalamic pituitary adrenal (HPA) Axis functioning and any medications that alter heart rate or skin conductance monitoring
16. Unable to follow the restrictions outlined in the protocol.
17. Legal status that would interfere with participation
18. Employed by the contract research organization (CRO) or are family members of the staff at the CRO
19. Previous participation in a cohort for any dose level of AEF0117.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs and SAEs as assessed by vital signs | since the first administration until 264 hours from last dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in vital signs
Incidence of treatment-emergent AEs and SAEs as assessed by ECGs | since the first administration until 264 hours from last dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in ECGs
Incidence of treatment-emergent AEs and SAEs as assessed by clinical laboratory values | since 24 hours from the first administration until 264 hours from last dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in clinical laboratory values from blood and urine samples.
Incidence of treatment-emergent AEs and SAEs as assessed by psychometric tests | 24 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in psychometric tests (Bond and Lader VAS, ARCI, POMS) and C-SSRS test.

SECONDARY OUTCOMES:
Pharmacokinetics of escalating multiple oral doses of AEF0117 | 264 hours from last dosing
  Peak Plasma Concentration (Cmax) induced by multiple doses of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating multiple oral doses of AEF0117 | 264 hours from last dosing
  Lowest Peak Plasma (Cmin) induced by multiple doses of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating multiple oral doses of AEF0117 | 264 hours from last dosing
  Time to maximum plasma concentration (tmax) of multiple doses of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating multiple oral doses of AEF0117 | 264 hours from last dosing
  Terminal elimination half-life (t1/2) based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating multiple oral doses of AEF0117 | 264 hours from last dosing
  Time to last measurable plasma concentration (tlast) based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating multiple oral doses of AEF0117 | 264 hours from last dosing
  Area under the plasma concentration versus time curve from time 0 (AUC0-t) based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacodynamics of escalating multiple oral doses of AEF0117 | 120 hours from last dosing
  Peak Plasma Concentration (Cmax) induced by multiple doses of AEF0117 on plasma pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.
Pharmacodynamics of escalating multiple oral doses of AEF0117 | 120 hours from last dosing
  Lowest Peak Plasma (Cmin) induced by multiple doses of AEF0117 on plasma pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.
Pharmacodynamics of escalating multiple oral doses of AEF0117 | 120 hours from last dosing
  Time to maximum plasma concentration (tmax) of multiple doses of AEF0117 on plasma pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.
Pharmacodynamics of escalating multiple oral doses of AEF0117 | 120 hours from last dosing
  Area under the plasma concentration versus time curve from time 0 (AUC0-t) of multiple doses of AEF0117 on plasma pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dobrow, MD, Principal Investigator — Biotrial Inc.
Locations (1):
- Biotrial Inc, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haney M, Vallee M, Fabre S, Collins Reed S, Zanese M, Campistron G, Arout CA, Foltin RW, Cooper ZD, Kearney-Ramos T, Metna M, Justinova Z, Schindler C, Hebert-Chatelain E, Bellocchio L, Cathala A, Bari A, Serrat R, Finlay DB, Caraci F, Redon B, Martin-Garcia E, Busquets-Garcia A, Matias I, Levin FR, Felpin FX, Simon N, Cota D, Spampinato U, Maldonado R, Shaham Y, Glass M, Thomsen LL, Mengel H, Marsicano G, Monlezun S, Revest JM, Piazza PV. Signaling-specific inhibition of the CB1 receptor for cannabis use disorder: phase 1 and phase 2a randomized trials. Nat Med. 2023 Jun;29(6):1487-1499. doi: 10.1038/s41591-023-02381-w. Epub 2023 Jun 8. PMID 37291212